CLINICAL TRIAL: NCT03340922
Title: MANual vs. automatIC Local Activation Time Annotation for Guiding Premature Ventricular Complex Ablation Procedures (MANIaC-PVC Study). A Randomized, Multicenter Study
Brief Title: MANual vs. automatIC Local Activation Time Annotation for Guiding Premature Ventricular Complex Ablation
Acronym: MANIaC-PVC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Principal Investigator, Centro Medico Teknon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Wavefront
Record Dates: First submitted 2017-11-03; First posted 2017-11-14 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Ventricular Premature Complexes; Catheter Ablation
Keywords: premature ventricular complex; catheter ablation; activation mapping; wavefront
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled and international multicenter study. All patients who fulfill the inclusion criteria will be consecutively enrolled and randomized on a 1:1 basis to each of the LAT annotation systems (WF vs. M-method) before the ablation procedure. Ablation will be directed to the earliest activation site identified with the assigned annotation system. Any change of the assigned annotation system during the procedure won't be allowed, thus being a reason for justifying study exclusion.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Automatic annotation of LAT (WF-method) (Experimental): The annotation of LAT in each acquired point will be automatically performed using the LAT annotation tool integrated into CARTO navigation system, called Wavefront (WF). Automatic annotation of LAT performed by the CARTO system uses the maximum negative slope of the distal U-EGM to set the timing of the mapping annotation, displayed on the corresponding B-EGM. Additionally, the automatic annotation of LAT will be aided by an ECG recognition pattern algorithm (included in the last version of CARTO), which is intended to avoid wrong annotation of ventricular complexes other than the clinical PVC.
  Interventions: Device: Automatic annotation of LAT (WF-method)
- Manual annotation of LAT (M-method) (Active Comparator): A detailed electrocardiogram (ECG)-gated activation map of the chamber of interest will be acquired using the CARTO navigation system. An experienced electrophysiologist will perform the annotation of LAT in each acquired point. The LAT will be measured from the onset of B-EGM (earliest positive or negative deflection) of the distal dipole of the mapping catheter to the defined reference. The use of the U-EGM as a guidance to identify the real onset of B-EGM will be decided under electrophysiologist criteria.
  Interventions: Device: Manual annotation of LAT (M-method)

INTERVENTIONS:
Device: Automatic annotation of LAT (WF-method) — Automatic annotation of LAT during PVC activation mapping. Acquisition of points will be automatically performed using the Wavefront (WF) annotation tool integrated into CARTO navigation system.
  Other Names: Wavefront
  Arms: Automatic annotation of LAT (WF-method)
Device: Manual annotation of LAT (M-method) — Conventional, manual annotation of LAT during PVC activation mapping. Acquisition of points will be performed using the CARTO navigation system by an expert electrophysiologist.
  Other Names: Manual
  Arms: Manual annotation of LAT (M-method)

SUMMARY:
Current navigation systems incorporate algorithms for automatic identification of local activation time (LAT). However, data about their utility and accuracy in premature ventricular complex (PVC) ablation procedures are scarce. This prospective, randomized study analyzes the accuracy and effectivity of an algorithmic method based on automatic annotation of the maximal negative slope of the unipolar electrogram within the window demarcated by the bipolar electrogram, compared with conventional, manual annotation during PVC ablation procedures.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled and international multicenter study. The investigators aim to analyze the accuracy of LAT annotation using a novel algorithmic method (Wavefront, CARTO, Biosense Webster, Diamond Bar, California, USA) (WF), based on automatic annotation of the maximal negative slope of the unipolar electrogram (U-EGM) within the window demarcated by the B-EGM, by comparison with conventional, manual annotation in a multicenter cohort of patients referred for PVC ablation. Further on, the automatic annotation of LAT will be aided by an ECG recognition pattern algorithm (included in the last version of CARTO), which is intended to avoid wrong annotation of ventricular complexes other than the clinical PVC. The investigators hypothesize that automatic LAT annotation (using WF and the ECG recognition algorithm) could be superior to conventional, manual annotation in terms of mapping success and could reduce both procedure time and radiofrequency time.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Indication for PVC ablation.
* Signed informed consent.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* PVC ablation procedures guided by pace-mapping (PASO® module); eg. low burden of PVCs during the study, mechanical impact during activation mapping.
* Impossibility to perform activation mapping with the required density of points in the region of interest (see section 4.5.3).
* Concomitant investigation treatments.
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Rates of mapping success, using the assigned mapping approach (automatic vs. manual), as defined in description | 12 months
  Mapping success will be defined as complete PVC abolition after RF applications at the earliest activation site (EAS) identified using the assigned mapping approach. A maximum of 2 RF applications with appropriate parameters (contact force, impedance drop, catheter stability) during a maximum of 45 seconds will be allowed. If the PVC is not abolished after 2 RF applications with appropriate parameters, mapping will not be considered successful.

SECONDARY OUTCOMES:
Mapping time | 12 months
Number of mapped chambers | 12 months
Accuracy of a proposed algorithm for selection of first chamber to map | 12 months
  In the case of PVCs arising from ventricular outflow tracts, we propose an algorithm to avoid subjective criteria, and to deal with eventual wrong selection of the first mapped chamber, leading to unnecessary RF applications. This algorithm involves a step-by-step analysis of the PVC-ECG morphology: precordial R/S transition and presence of one or more of the following clinical items, which have been previously related with a left origin: male gender, hypertension, or age > 50 years.
Number of target points | 12 months
  Target point is defined as any suspected PVC-site of origin where RF is delivered according to mapping data. Therefore, for one case there can be found a single target point with multiple RF applications, or multiple target points with one single RF application. The maximum distance between 2 RF applications to be considered at the same target point will be defined as 5 mm (equivalent to a 1-cm2 area).
Radiofrequency (RF) time | 12 months
Number of RF applications | 12 months
Acute procedure success | 12 months
  Complete elimination of the PVC at the end of the procedure.
Clinical success | 1 month
  Reduction of, at least, 80% in the 24-hour PVC burden 1 month after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Berruezo, MD, PhD, Principal Investigator — Centro Medico Teknon; Felipe Bisbal, MD, PhD, Principal Investigator — Hospital Universitari German Trias i Pujol (Badalona, Spain); Alonso Pedrote, MD, PhD, Principal Investigator — Virgen del Rocio University Hospital (Sevilla, Spain); Diego Penela, MD, PhD, Principal Investigator — Ospedale Guglielmo da Saliceto (Piacenza, Italy); Juan Fernández-Armenta, MD, PhD, Principal Investigator — Puerta del Mar University Hospital (Cadiz, Spain)
Locations (1):
- Antonio Berruezo, MD, PhD, Barcelona, Spain

REFERENCES:
- [Background] Stevenson WG, Soejima K. Recording techniques for clinical electrophysiology. J Cardiovasc Electrophysiol. 2005 Sep;16(9):1017-22. doi: 10.1111/j.1540-8167.2005.50155.x. PMID 16174026
- [Background] Liuba I, Walfridsson H. Activation mapping of focal atrial tachycardia: the impact of the method for estimating activation time. J Interv Card Electrophysiol. 2009 Dec;26(3):169-80. doi: 10.1007/s10840-009-9437-0. Epub 2009 Oct 29. PMID 19866350
- [Background] Ndrepepa G, Caref EB, Yin H, el-Sherif N, Restivo M. Activation time determination by high-resolution unipolar and bipolar extracellular electrograms in the canine heart. J Cardiovasc Electrophysiol. 1995 Mar;6(3):174-88. doi: 10.1111/j.1540-8167.1995.tb00769.x. PMID 7620643
- [Background] El Haddad M, Houben R, Stroobandt R, Van Heuverswyn F, Tavernier R, Duytschaever M. Novel algorithmic methods in mapping of atrial and ventricular tachycardia. Circ Arrhythm Electrophysiol. 2014 Jun;7(3):463-72. doi: 10.1161/CIRCEP.113.000833. Epub 2014 May 14. PMID 24829224
- [Background] Andreu D, Berruezo A, Fernandez-Armenta J, Herczku C, Borras R, Ortiz-Perez JT, Mont L, Brugada J. Displacement of the target ablation site and ventricles during premature ventricular contractions: relevance for radiofrequency catheter ablation. Heart Rhythm. 2012 Jul;9(7):1050-7. doi: 10.1016/j.hrthm.2012.02.018. Epub 2012 Feb 15. PMID 22342861
- [Background] Penela D, De Riva M, Herczku C, Catto V, Pala S, Fernandez-Armenta J, Acosta J, Cipolletta L, Andreu D, Borras R, Rios J, Mont L, Brugada J, Carbucicchio C, Zeppenfeld K, Berruezo A. An easy-to-use, operator-independent, clinical model to predict the left vs. right ventricular outflow tract origin of ventricular arrhythmias. Europace. 2015 Jul;17(7):1122-8. doi: 10.1093/europace/euu373. Epub 2015 Feb 10. PMID 25672982
- [Background] Penela D, Van Huls Van Taxis C, Van Huls Vans Taxis C, Aguinaga L, Fernandez-Armenta J, Mont L, Castel MA, Heras M, Tolosana JM, Sitges M, Ordonez A, Brugada J, Zeppenfeld K, Berruezo A. Neurohormonal, structural, and functional recovery pattern after premature ventricular complex ablation is independent of structural heart disease status in patients with depressed left ventricular ejection fraction: a prospective multicenter study. J Am Coll Cardiol. 2013 Sep 24;62(13):1195-202. doi: 10.1016/j.jacc.2013.06.012. Epub 2013 Jul 10. PMID 23850913

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT03340922/Prot_SAP_000.pdf